CLINICAL TRIAL: NCT02720003
Title: A Prospective, Multicenter, Single Arm Trial Evaluating the BARD Lutonix Drug-Coated Balloon (LTX DCB) for Treatment of Femoropopliteal Arteries (LEVANT China)
Brief Title: A Single Arm Trial Evaluating the BARD Lutonix Drug-Coated Balloon (LTX DCB) for Treatment of Femoropopliteal Arteries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC1401PV
Record Dates: First submitted 2016-02-26; First posted 2016-03-25 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Femoral Artery Stenosis; Femoral Artery Occlusion; Stenosis of Popliteal Arteries; Occlusion of Popliteal Arteries
Keywords: Atherosclerosis; Superficial Femoral Artery; Proximal Popliteal Artery
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LTX DCB (Experimental): Patients treated with Bard Lutonix DCB
  Interventions: Device: LTX DCB

INTERVENTIONS:
Device: LTX DCB — Treatment with a drug-coated balloon

SUMMARY:
To assess the safety and efficacy of the BARD LTX DCB for treatment of stenosis or occlusion of the superficial femoral and popliteal arteries.

DETAILED DESCRIPTION:
The study will enroll patients presenting with claudication or ischemic rest pain due to stenotic lesions in the superficial femoral or popliteal artery and a patent outflow artery to the foot. After successful pre-dilatation, subjects determined by the investigator not to require stenting based on defined angiographic criteria will receive the BARD LTX DCB. .

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and < 85 years of age;
* Documented diagnosis of peripheral arterial disease (PAD) with Rutherford Classification stages 2-4;
* Patient is willing to provide informed consent and comply with the required - follow up visits, testing schedule and medication regimen;

Angiographic Criteria

* Single lesion or up to two focal lesions (not separated by >3 cm) (total vessel segment length ≤20 cm) in native superficial femoral and/or popliteal arteries;
* ≥70% diameter stenosis by visual estimate;
* Lesion location starts ≥1 cm below the common femoral bifurcation and terminates distally ≤2 cm below the tibial plateau AND ≥1 cm above the origin of the TP trunk;
* De novo lesion(s) or non-stented restenotic lesion(s) >90 days from prior angioplasty procedure;
* Lesion is located at least 3 cm from any stent, if target vessel was previously stented;
* Target vessel diameter between ≥4 and ≤7 mm and able to be treated with available device size matrix;
* Successful, uncomplicated (without use of a crossing device) antegrade wire crossing of lesion;
* A patent inflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of inflow iliac and/or common femoral artery lesions);
* No vascular interventions, surgical or interventional procedures within 2 weeks before and/or planned 30 days after the protocol treatment.

Exclusion Criteria

Patients will be excluded if ANY of the following conditions apply:

* Breastfeeding or pregnant or planning on becoming pregnant or men intending to father children;
* Life expectancy of < 2 year;
* Patient is currently participating in an investigational drug or other device study or previously enrolled in this study;
* History of stroke within 3 months;
* History of MI, thrombolysis or angina within 2 weeks of enrollment;
* Renal failure or chronic kidney disease with MDRD GFR ≤30 ml/min per 1.73 m2 (or serum creatinine ≥2.5 mg/dL within 30 days of index procedure or treated with dialysis);
* Diagnosed active systemic infection or uncontrolled coagulopathy within 14 days prior to index procedure
* Prior vascular surgery of the index limb, with the exception of remote common femoral patch angioplasty separated by at least 2 cm from the target lesion;
* Inability to take required study medications or allergy to paclitaxel or paclitaxel related compounds or contrast that cannot be adequately managed with pre- and post-procedure medication;
* The lesion is a post-DCB restenosis, or within or adjacent to an aneurysm; Ipsilateral retrograde access;
* There is no normal proximal arterial segment in which duplex flow velocity can be measured;
* Known inadequate distal outflow (≥50% stenosis of distal popliteal and/or all three tibial vessels;), or planned future treatment of vascular disease distal to the target lesion;
* Sudden symptom onset, acute vessel occlusion, or acute or sub-acute thrombus in target vessel;
* Severe calcification that renders the lesion un-dilatable or failed pre-dilatation, defined by a residual stenosis >50% or major flow limiting dissection;
* Use of adjunctive treatment modalities (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, embolic protection device, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-03; Primary Completion 2018-10 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy - Percentage of Subjects With Primary Patency of the Target Lesion at One Year | 0-12 months
  Primary Patency is defined as the absence of target lesion restenosis (defined by DUS peak systolic velocity ratio [PSVR] ≥2.5 and/or abnormal waveforms, as determined by an Independent Core Laboratory) and freedom from target lesion revascularization (TLR).
Primary Safety - Percentage of Subjects With Composite of Freedom From All-cause Peri-operative Death and Freedom From the Following: Index Limb Amputation, Index Limb Re-intervention, and Index-limb-related Death | 0-30 days
  Primary Safety - Percentage of Subjects With Composite of Freedom From All-cause Peri-operative Death and Freedom From the Following: Index Limb Amputation, Index Limb Re-intervention, and Index-limb-related Death

SECONDARY OUTCOMES:
Device Success | 1 month
Technical Success | 1 month
Acute Technical Success | 1 month
Procedural Success | 1 month
Percentage of Subjects with Primary Patency of the Target Lesion | 24 months
Target Lesion Revascularization | 24 months
  Proportion of subjects with target lesion revascularization through 24 months
Change in Rutherford Classification | 24 months
  Mean change in Rutherford Classification from baseline through 24 months
Change in Ankle Brachial Index | 24 months
  Mean change in ankle brachial index from baseline through 24 months
Percentage of subjects who died from any cause | 24 months
Amputation-free Survival | 24 months
  Percentage of subjects with above-the-ankle amputation-free survival
Percentage of subjects with Target Vessel Revascularization | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Professor, Principal Investigator — Chinese PLA General Hospital; Weiguo Fu, Professor, Principal Investigator — Fudan University; Fuxian Zhang, Principal Investigator — Beijing Shijitan Hospital. CMU; Tong Qiao, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Lan Zhang, Principal Investigator — RenJi Hospital; Xinwu Lu, Principal Investigator — Shanghai Ninth People's Hosptial , Shanghai JiaoTong University School of Medicine; Feng Wang, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Pingfan Guo, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Shaomang Lin, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University; Wei Bi, Principal Investigator — The Second Hospital of Hebei Medical University; Jichun Zhao, Principal Investigator — West China Hospital; Jianjun Jiang, Principal Investigator — Qilu Hospital of Shandong University; Haofu Wang, Principal Investigator — The Affiliated Hospital of Qingdao University; Xiangchen Dai, Principal Investigator — Tianjin Medical University General Hospital
Locations (14):
- China (14):
  - Beijing Shijitan Hospital. CMU, Beijing, Beijing Municipality
  - Chinese- PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanjing Drum Tower Hospital,The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Ninth People's Hosptial , Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - RENJI Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - General Hospital of Tianjin Medical University, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided